CLINICAL TRIAL: NCT02102087
Title: A Matched, Open Label Study to Evaluate the Effectiveness of the MMT Initial Specimen Diversion Device in Reducing Blood Culture Contamination When Compared to Laboratory Standard Procedures
Brief Title: Study to Evaluate the Effectiveness of the Initial Specimen Diversion Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magnolia Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMT1302
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Septicemia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial Specimen Diversion Device (ISDD) (Experimental): The ISDD will be used in conjunction with standard blood culture bottles.
  Interventions: Device: Initial Specimen Diversion Device (ISDD)
- Lab standard practice (LSP) (Active Comparator): A standard blood culture kit will be used.
  Interventions: Device: Lab standard practice (LSP)

INTERVENTIONS:
Device: Initial Specimen Diversion Device (ISDD)
  Arms: Initial Specimen Diversion Device (ISDD)
Device: Lab standard practice (LSP)
  Arms: Lab standard practice (LSP)

SUMMARY:
This is a matched, open label study to evaluate the Initial Specimen Diversion Device (ISDD) in reducing the contamination rate in blood culture analysis. Blood culture data will be derived from inpatient and/or outpatient settings in a variety of hospital departments (e.g. ER, surgical, medical, etc.). Only samples that are collected via peripheral venipuncture may be included in this study. The ISDD will be compared to current laboratory practices for the collection of blood for culture purposes. Laboratory Standard Procedures (LSP) is defined as collection of venipuncture blood for culture without an initial diversion method to divert and sequester potential blood contaminants.

ELIGIBILITY:
Inclusion Criteria:

* Adults >19 years old

Exclusion Criteria:

* Not a good candidate for direct-to-media (DTM) technique

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of blood culture contamination when using the Initial Specimen Diversion Device (ISDD) compared to Laboratory Standard Procedures (LSP) | Baseline
  Comparison of contamination for each clinical episode. The proportions of discordant contamination episodes will be compared between the Initial Specimen Diversion Device and Lab Standard Practice using McNemar's test.

SECONDARY OUTCOMES:
Occurrence rate of adverse device effects | Baseline
  As the device under study enhances the blood diversion procedure during blood culture collection, and is part of standard blood collection standards, adverse device effects are not expected as a result of use of this device, but shall be recorded consistent with the adverse event definitions found in 21 CFR 812. As this is a commercially available device, medical device reporting shall be performed in accordance with 21 CFR 803, as applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Rupp ME, Cavalieri RJ, Marolf C, Lyden E. Reduction in Blood Culture Contamination Through Use of Initial Specimen Diversion Device. Clin Infect Dis. 2017 Jul 15;65(2):201-205. doi: 10.1093/cid/cix304. PMID 28379370